CLINICAL TRIAL: NCT07062146
Title: Evaluation of the Effect of Reiki on Pain After Spinal Fusion: A Comparative, Randomized, Pilot Study
Brief Title: Evaluation of the Effect of Reiki on Pain After Spinal Fusion
Acronym: REDAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Bizet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2024-A02685-42
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Chirurgical Intervention
MeSH Terms: interventions — Therapeutic Touch; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard treatment (analgesic + kinesitherapy sessions) + Treatment session (Reiki) (Experimental): treatment with reiki session
  Interventions: Other: reiki
- standard treatment (analgesic + kinesitherapy sessions) + Treatment session (Sham) (Placebo Comparator): treatment with sham session
  Interventions: Other: Sham (No Treatment)

INTERVENTIONS:
Other: reiki — Reiki sessions for 30 minutes, on Day-7 before the surgery and on D15 after the surgery
  Arms: standard treatment (analgesic + kinesitherapy sessions) + Treatment session (Reiki)
Other: Sham (No Treatment) — Sham sessions for 30 minutes, on D-7 before the surgery and on D15 after the surgery,
  Arms: standard treatment (analgesic + kinesitherapy sessions) + Treatment session (Sham)

SUMMARY:
This study involves patients undergoing lumbar spine surgery (lumbar arthrodesis). It compares the effects of Reiki, an energy-based therapy, with conventional approaches to relieve postoperative pain.

The goal is to determine whether this non-drug method can help reduce pain, limit the use of painkillers, and enhance patient comfort during recovery.

ELIGIBILITY:
Inclusion Criteria:

* - Subject aged 18 years or older;
* Referred for a lumbar fusion of up to 3 levels.
* Absence of participation in another clinical study.
* Subject affiliated with a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Neuropathic patient
* Presence of neuropathic pain
* Diagnosis of fibromyalgia
* Received therapeutic touch, polarity therapy, or professional massage therapy in the past four weeks
* Unable to undergo medical follow-up for the study
* Adult subject protected by law, under guardianship or trusteeship

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
pain will be assessed at Day 15 using the VAS ( Visial Analog Scale) | DAY 15
  The Visual Analog Scale is a subjective measurement tool commonly used to assess the intensity of pain. It consists of a horizontal 10-centimeter line on which the patient marks a point that reflects their experience.
  Minimum and maximum values:
  0 = complete absence of the symptom
  10 = the most severe imaginable intensity of the symptom
  Score interpretation:
  Higher scores indicate greater symptom intensity
  Lower scores indicate lesser intensity

SECONDARY OUTCOMES:
Quality of life will be assessed using the SF12 | DAY 30
  The SF-12 (Short-Form Health Survey) a validated questionnaire designed to assess health-related quality of life across physical and mental domains. It is a shortened version of the SF-36, containing 12 items that cover eight key health dimensions.
  Scoring:
  * Higher scores indicate better health status in each domain
  * Each item uses Likert-type responses ("Excellent" to "Poor", or "All of the time" to "None of the time")
Daily pain intensity will be reported | from Day 1 to Day 30
  This daily diary was designed by the research team to record pain intensity using the Visual Analog Scale (VAS), from the day of discharge up to 30 days post-intervention.
  The Visual Analog Scale is a subjective measurement tool commonly used to assess the intensity of pain. It consists of a horizontal 10-centimeter line on which the patient marks a point that reflects their experience.
  * Minimum and maximum values:
    0 = complete absence of the symptom 10 = the most severe imaginable intensity of the symptom
  * Score interpretation:
  Higher scores indicate greater symptom intensity Lower scores indicate lesser intensity
evaluation of patient's overall satisfaction and treatment response | at Day 30
  the Clinical Global Impression (CGI) is a clinician-rated scale used to assess the global change in a patient's condition following a medical or therapeutic intervention, compared to their state at baseline.
  Evaluated on a 7-point scale :
  1. = Very much improved
  2. = Much improved
  3. = Minimally improved
  4. = No change
  5. = Minimally worse
  6. = Much worse
  7. = Very much worse
Assessment of the condition of the scar at the lumbar level | at Day 15 and Day 30
  The International Visual Wound Color Scale (IVWCS) This scale is a visual assessment tool that helps clinicians evaluate wound healing by identifying and interpreting the dominant colors present in the wound bed.
  Each color corresponds to a specific tissue type or healing stage.
  Color Categories and Their Meanings:
  * Red: Indicates healthy granulation tissue, which is essential for wound repair. Suggests active healing and good blood supply Requires protection and monitoring for infection
  * Yellow: Often associated with slough or exudate, which may signal infection or delayed healing.
  Requires cleaning and possibly debridement May indicate microbial presence or inflammation
  - Black: Represents necrotic tissue (dead tissue), often due to poor blood supply.
  Requires urgent medical attention Typically treated with debridement and moist dressings
antalgic consumption will be reported | from day 1 to day 30
  This daily diary was designed by the research team and records the daily consumption of analgesics from the day of discharge to 30 days post-intervention.
  Classification of Analgesics in the Daily Diary Analgesic consumption will be categorized according to the standard analgesic step classification:
  * Step 1: Non-opioid analgesics (paracetamol, NSAIDs)
  * Step 2: Weak opioids (codeine, tramadol)
  * Step 3: Strong opioids (morphine, fentanyl)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Bizet, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided